

## FREE AND CLARIFIED CONSENT

This is a consent form to participate in the research entitled: "Strength and Muscle Activation of Runners Quadriceps After 8 Weeks of Intervention With Elastic Bandage"

This information is being provided for your voluntary participation in this study, which aims to investigate the effect of elastic bandage on the peak isokinetic torque of knee flexors and extensors and surface electromyography in runners.

The objective of this research is to evaluate, in the long term, the influenced elastic bandage in the gain of muscular strength of the quadriceps through the peak isokinetic torque (muscle strength) of knee flexors and extensors and surface electromyography (electrical activity of the muscle) of the rectus femoris.

You will participate in two assessments, one before and one after the interventions, involving tests of muscle strength and surface electromyography using gold standard assessment instruments (isokinetic and electromyograph). The results of the study may be published in magazines, books, or scientific events, which will keep your identity confidential, the data collected will be used only for educational and research purposes. The study was approved by the Ethics and Research Committee CEP - UNOPAR under No. 3,059,113, in compliance with the provisions of resolution 466/12 of the National Health Council.

The entire procedure will be based on the literature on the topic, in addition to respecting your individuality. This study will be important to expand knowledge about the techniques used. The risks to which the volunteers will be submitted will be minimal and may include: musculoskeletal discomforts after evaluation and allergies to elastic bandages. This study will assess the level of muscle strength and muscle activation before and after 8 weeks of running training, providing participants with the result of their assessments in order to encourage them to improve their performance.

The interventions will be carried out by a student in the PhD course in Rehabilitation Science, from UEL-UNOPAR. Questions related to the procedures of this study should be addressed to the person responsible for the same, by calling: (43) 9 9172 2201 at the Health Sciences Center (CCS) of the State University of Northern Paraná (UENP).

You are not required to participate in this study and can withdraw during the study at any time, without any loss. As a result, there are no personal expenses on your part to participate in this study. Just as there is no financial compensation. If you voluntarily agree to participate in this study, you must sign this document in the presence of a witness.

| Volunteer signature | Date: <u>///</u> |
|---|---|
| Witness signature | Date: / / |
| Inappropriately obtained the Free and Informed Con | nsent of this volunteer to participate in this study. |
| Researcher's signature | Date: / / |